CLINICAL TRIAL: NCT00872950
Title: Open Label Trial Of 3,4-Diaminopyridine In Lambert-Eaton Myasthenic Syndrome (LEMS) and Congenital Myasthenic Syndromes (CMS)
Brief Title: 3,4-Diaminopyridine Use in Lambert-Eaton Myasthenic Syndrome(LEMS) and Congenital Myasthenic Syndromes (CMS)
Acronym: LEMS
Status: Approved for marketing | Type: Expanded Access
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2001-040
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Lambert-Eaton Myasthenic Syndrome; Congenital Myasthenic Syndrome
Keywords: LEMS; CMS; 3,4 DIAMINOPYRIDINE; 3,4 DAP
MeSH Terms: conditions — Lambert-Eaton Myasthenic Syndrome; Myasthenic Syndromes, Congenital | interventions — Amifampridine

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: 3,4-DIAMINOPYRIDINE — Treatment will begin with a low dose and will be increased as clinically needed as tolerated. The upper limit will be a total of 100mg/day.
  Other Names: 3,4 DAP

SUMMARY:
The purpose of this study is to determine the effectiveness and adverse effects of 3,4-diaminopyridine for the treatment of the Lambert-Eaton Myasthenic Syndrome (LEMS) and Congenital Myasthenic Syndromes (CMS).

DETAILED DESCRIPTION:
This is an open-label, non-randomized, non-comparative expanded access study. Up to 25 patients with clinically proven paraneoplastic or primary autoimmune LEMS per EMG and positive voltage-gated calcium channel antibody serology, OR patients with clinically proven CMS per electromyogram (EMG), biopsy or genetic testing who meet the selection criteria outlined in sections 3.1 and 3.2 will be enrolled in this study. Subjects will receive 3,4-diaminopyridine (3,4-DAP) starting with a low dose and titrating up per efficacy and patient tolerance to a maximum daily dose of 100mg . Treatment will continue until the subject experiences a treatment-limiting toxicity, voluntarily withdraws consent, transfers to another site, dies, becomes lost to follow-up, is no longer receiving clinical benefit from 3,4-DAP (in the opinion of the subject and/or the investigator), or the Jacobus Pharmaceuticals or the FDA discontinues the study.

ELIGIBILITY:
Inclusion Criteria:

* LEMS diagnosis OR Pre or Post Synaptic CMS diagnosis
* 18 years or older
* Females must have negative pregnancy test and be willing to practice an effective form of birth control
* No prolonged QT syndrome as indicated by baseline EKG

Exclusion Criteria:

* Known sensitivity to 3,4-DIAMINOPYRIDINE
* History of seizures and/or severe asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jayashri Srinivasan, MD,MCRP,PhD, Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Hospital & Medical Center, Burlington, Massachusetts, United States

REFERENCES:
- See also: Lahey Hospital & Medical Center — http://www.lahey.org